CLINICAL TRIAL: NCT05680311
Title: Is Autotaxin a Promising Biomarker for Breast Cancer
Brief Title: Autotaxin: a Potential Biomarker for Breast Cancer.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Etlik City Hospital (Other Government)
Collaborators: Diskapi Yildirim Beyazit Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Gaye Seker, Assistant Professor of Surgery, Ankara Etlik City Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: autotaxin1
Record Dates: First submitted 2022-12-26; First posted 2023-01-11 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Breast Cancer
Keywords: breast cancer; autotaxin; tumor marker
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Breast Cancer Patients (Active Comparator): Group of patients with verified breast cancer diagnosis
  Interventions: Biological: measurement of serum autotaxin serum level
- Non-Cancer patients (Sham Comparator): Group of healthy patients with no verified any type of cancer.
  Interventions: Biological: measurement of serum autotaxin serum level

INTERVENTIONS:
Biological: measurement of serum autotaxin serum level — autotaxin expression

SUMMARY:
The goal of this clinical trial is to test the efficiency of Autotaxin (ATX) as a biomarker for breast cancer patients.

The main questions it aims to answer are;

* is ATX a reliable tumor marker for breast cancer patients in diagnosis
* can ATX differentiate cancer patients from non-cancer ones

DETAILED DESCRIPTION:
80 breast cancer patients and 30 normal patients with no known cancer history were enrolled in this study. All patients were female. The mean ages of cancer patients were 58.2 and 52.7 consecutively for cancer and non-cancer patients. The mean serum ATX levels of cancer and non-cancer patients were 1570.72 and 121.86 ng/mL consecutively (p=0.001). The cut-off value of ATX serum level was 178.49ng/mL according to the ROC analysis. The area under the ROC curve was 0.901showing that ATX is very efficient in distinguishing between two diagnostic groups (diseased/normal). ATX also showed good correlations with known tumor markers (CEA, CA15-3, CA125 levels). ATX levels were still higher than the cut-off value even in cancer patients with normal or low classical tumor marker levels.

ELIGIBILITY:
Inclusion Criteria:

* Preoperatively diagnosed breast cancer patients with no synchronous cancer and without known hepatic or other inflammatory disorders.

Exclusion Criteria:

* Patients with benign breast diseases and no known cancer history.

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-03-15 (Actual)

PRIMARY OUTCOMES:
Autotaxin as a tumor marker | preoperative period
  Diagnostic value of Autotaxin in breast cancer

CONTACTS AND LOCATIONS:
Overall Officials: Duray Seker, Professor, Study Chair — Ankara Etlik City Hospital
Locations (1):
- Ankara Etlik City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD
Supporting Information: Study Protocol
Time Frame: from the onset of publication
Access Criteria: Only access criteria is citing the article

REFERENCES:
- [Result] Lukasiewicz S, Czeczelewski M, Forma A, Baj J, Sitarz R, Stanislawek A. Breast Cancer-Epidemiology, Risk Factors, Classification, Prognostic Markers, and Current Treatment Strategies-An Updated Review. Cancers (Basel). 2021 Aug 25;13(17):4287. doi: 10.3390/cancers13174287. PMID 34503097
- [Result] Gaetano CG, Samadi N, Tomsig JL, Macdonald TL, Lynch KR, Brindley DN. Inhibition of autotaxin production or activity blocks lysophosphatidylcholine-induced migration of human breast cancer and melanoma cells. Mol Carcinog. 2009 Sep;48(9):801-9. doi: 10.1002/mc.20524. PMID 19204929
- [Result] Brindley DN, Tang X, Meng G, Benesch MGK. Role of Adipose Tissue-Derived Autotaxin, Lysophosphatidate Signaling, and Inflammation in the Progression and Treatment of Breast Cancer. Int J Mol Sci. 2020 Aug 18;21(16):5938. doi: 10.3390/ijms21165938. PMID 32824846